CLINICAL TRIAL: NCT02572375
Title: An Open-Label, Randomized, Multiple-Dose, 2-Way Crossover Comparative Bioavailability Steady State Study of Codeine Phosphate/Guaifenesin Extended-Release Tablet in Healthy Subjects
Brief Title: Codeine Phosphate/Guaifenesin ER Tablet 30 mg/600 mg Steady State Clinical Study
Acronym: COGUSS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nexgen Pharma, Inc (Industry)
Collaborators: Pharmaceutical Research Unit, Jordan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: COGU510
Record Dates: First submitted 2015-04-14; First posted 2015-10-08 (Estimated); Last update posted 2017-03-29 (Actual); Status verified 2017-03

CONDITIONS: Cough
MeSH Terms: conditions — Cough | interventions — Codeine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Codeine Phosphate/Guaifenesin ER Tablet (Experimental): Patients receiving an extended release tablet dosage form of a combination drug of Codeine Phosphate and Guaifenesin twice a day for 6 and a half days total. Total dosage [2 tablets] is 60 mg Codeine Phosphate and 1200 mg Guaifenesin twice a day for a daily total of 120 mg Codeine Phosphate and 2400 mg Guaifenesin.
  Interventions: Drug: Codeine Phosphate/Guaifenesin ER Tablet
- Codeine Phosphate/Guaifenesin IR Tablet (Active Comparator): Patients receiving an immediate release tablet dosage form of a combination drug of Codeine Phosphate and Guaifenesin six times a day for 6 and a half days total. Dosage is 20 mg Codeine Phosphate and 400 mg Guaifenesin six times a day for a daily total of 120 mg Codeine Phosphate and 2400 mg Guaifenesin.
  Interventions: Drug: Codeine Phosphate/Guaifenesin IR Tablet

INTERVENTIONS:
Drug: Codeine Phosphate/Guaifenesin ER Tablet — Provide two Codeine Phosphate and Guaifenesin ER Tablet every 12 hours for 6 1/2 days.
  Other Names: Lot 100171
  Arms: Codeine Phosphate/Guaifenesin ER Tablet
Drug: Codeine Phosphate/Guaifenesin IR Tablet — Provide one Codeine Phosphate and Guaifenesin IR Tablet every 4 hours for 6 1/2 days
  Other Names: Lot 100168
  Arms: Codeine Phosphate/Guaifenesin IR Tablet

SUMMARY:
The objectives of this pivotal study are:

1. to evaluate bioavailability of an extended-release and immediate release Codeine Phosphate/Guaifenesin tablet at steady state following multiple oral administration
2. to assess the safety and tolerability of this Codeine Phosphate/Guaifenesin extended release formulation.

DETAILED DESCRIPTION:
This study will be a single-center, Two-site open-label, randomized, multiple-dose, two-treatment, two-period crossover design. During the course of the study, thirty eight (38) healthy adult volunteers will receive multiple doses of Codeine Phosphate/ Guaifenesin extended-release tablet 30 mg/600 mg and multiple doses of an IR Codeine Phosphate/ Guaifenesin immediate-release tablet 20 mg/400 mg tablet in two separate treatment periods.

Volunteers will enter the clinic the day prior [approximately 12 hours] to each dosing and will be confined in the clinic for 7 nights for each treatment period. The extended release tablet (test) will be administered as two tablets two times a day, 12 hours apart, and the immediate release tablet (reference) will be administered as one tablet six times a day, 4 hours apart. Pre-dose blood samples will be collected prior to morning dose on Days 1, 2, 3, 4, 5, 6 and 7. On Day 7, Two extended release tablets will be given once in the morning and the immediate release tablet will be given three times, in the morning and 4 and 8 hours later. Serial blood samples will be collected on Day 7 for up to 12 hours post morning dose.

On Day 7 volunteers will be released from the study site after the 12-hour blood collection if clinically appropriate and will return to the study site to start the next treatment after a minimum of 7 days of wash-out period, which begins the morning after the last dose taken of the previous Period.

ELIGIBILITY:
Inclusion Criteria:

* Healthy non-smoking volunteers (Female volunteers on a stable contraceptive medication regimen (> 3 months) may continue during the course of the study but its use must be documented), 18 to 45 years of age, inclusive; Ethnic Group: Arab & Mediterranean.

  * Race: Mixed skin (white & black skin people).
  * Body Mass Index (BMI) between 18 and 32 kg/m2, inclusive (minimum of 50 kg weight);
  * willing and able to comply with the appropriate instructions necessary to complete the study, and;
  * Fully informed of the risks of entering the study and willing to provide written informed consent.
  * Subject is available for the whole study period and gave written informed consent
  * If female, must be practicing abstinence or using a medically acceptable form of contraception (e.g., intrauterine device, hormonal birth control [continuously used for at least 3 months before first dose], or double barrier method). For the purpose of this study, all females are considered to be of childbearing potential unless they have been post - menopausal, biologically sterile, or surgically sterile (i.e., hysterectomy, bilateral oophorectomy, or tubal ligation) for more than one (1) year
  * Normal Physical examination.
  * Vital signs within normal ranges.
  * All laboratory screening results within the normal range, or being assessed as clinically Non-significant by the attending physician.
  * Normal Kidney and Liver functions test.

Exclusion Criteria:

* • Women of childbearing potential who don't use any contraceptive method, pregnant and/or lactating women.

  * Ethnic Group (Non- Arab &/ or Non- Mediterranean)
  * A significant abnormality in the pre-study physical examination that would place the volunteer at risk during participation in the trial;
  * A clinical laboratory test value outside of the accepted reference range that is deemed by the Investigator to be clinically significant;
  * Require prescription medication on a regular basis;
  * A clinically significant illness during the 28 days prior to Period 1 dosing (as determined by the Investigator);
  * History of serious illness that can impact fate of drugs
  * History of gastrointestinal obstruction, constipation, inflammatory bowel disease, gallbladder disease, pancreas disorder over last 2 years, or recent (over last 3 years) gastrointestinal tract surgery, including gall bladder resection;
  * Known history or presence of cardiac, pulmonary, endocrine, musculoskeletal, neurological, hematological or disease.
  * Subjects with acute pulmonary insufficiency, respiratory depression, acute or chronic severe respiratory insufficiency or history of any of these
  * History of head injury, seizures over last 4 years deemed by the Investigator to be clinically significant;
  * Mental disease
  * History of kidney disease or urination problem over last 2 years deemed by the Investigator to be clinically significant
  * Subjects with renal and/or hepatic insufficiency should be excluded
  * Presence of any significant physical or organ abnormality
  * History of low blood pressure is deemed by the Investigator to be clinically significant;
  * A positive Hepatitis B surface antigen, Hepatitis C antibody screen, or a reactive HIV antibody screen;
  * Known or suspected hypersensitivities, allergies, or other contraindications to Codeine or a related opioid and/or Guaifenesin;
  * History of severe allergy or allergic reactions to study drug or related drugs or heparin
  * Known history or presence of food allergies, or any condition known to interfere with the absorption, distribution, metabolism or excretion of drugs
  * Known or suspected history of drug abuse within lifetime as judged by the Investigator;
  * History of alcohol abuse or excessive intake of alcohol within last 5 years as judged by the Investigator;
  * Positive screen for drugs of abuse, alcohol, or cotinine (nicotine) at screening or on admission to the unit prior to administration of investigational products;
  * Use of drugs that induce or inhibit the hepatic metabolizing cytochrome P450 2D6 enzymes, within 30 days prior to administration of study formulations. Examples of inducers include: piperidins, carbamazepine, dexamethasone, rifampin. Examples of inhibitors include: cimetidine, diphenhydramine, fluvastatine, methadone, and ranitidine;
  * Use of prescription medications within 21 days and OTC medications (including vitamins or herbal products) within 7 days (excluding flu vaccination) prior to the first administration of the study medication without Sponsor approval;
  * Intake of Alcohol 48 before each study drug administration, and caffeine, or xanthine beverages 24 hrs before each study drug administration.
  * Use of any investigational drug within 30 days prior to first dosing;
  * Use of any tobacco-containing product within 6 months of first dosing;
  * Donated more than 400 mL of blood within 4 weeks before first dosing;
  * Participation in another bioequivalence study and/or Clinical trials within 80 days prior to the start of this study Period I
  * Exhausting physical exercise in the last 48 hours (e.g. weight lifting) or any recent significant change in dietary or exercise habits.
  * Abnormal vital signs
  * Abnormal Kidney and Liver functions test.
  * In the opinion of the Investigator, unlikely or unable to successfully complete the study;
  * Volunteer is vegetarian.
  * Vomiting, Diarrhea on admission.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2014-10; Primary Completion 2014-11 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Peak Plasma Concentration (Cmax) | One week
  Determination peak plasma concentration of each active ingredient during 12 hours following six days of dosing
Area under the plasma concentration versus time curve (AUC) | One week
  Determination of total area under the plasma concentration versus time curve (AUC) during the 12 hours following 6 days of dosing.

CONTACTS AND LOCATIONS:
Overall Officials: Rana T Bustami, PhD, Principal Investigator — Pharmaceutical Research Unit, Jordan
Locations (1):
- Pharmaceutical Research Unit, Amman, Jordan